CLINICAL TRIAL: NCT00002465
Title: Phase I/II Study of High-Dose Megestrol in Breast or Endometrial Carcinoma or Mesothelioma
Brief Title: High-Dose Megestrol in Treating Patients With Metastatic Breast Cancer, Endometrial Cancer, or Mesothelioma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Vincent Medical Center - Los Angeles (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000076422; SVMC-V89-0296; NCI-V89-0296
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-07

CONDITIONS: Breast Cancer; Endometrial Cancer; Malignant Mesothelioma
Keywords: stage IV breast cancer; recurrent breast cancer; advanced malignant mesothelioma; recurrent malignant mesothelioma; stage IV endometrial carcinoma; recurrent endometrial carcinoma
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Mesothelioma, Malignant | interventions — Megestrol Acetate

INTERVENTIONS:
Drug: megestrol acetate

SUMMARY:
RATIONALE: Some hormones can stimulate the growth of some types of cancer cells. Hormone therapy using megestrol may fight cancer by reducing the production of these hormones.

PURPOSE: Phase I/II trial to study the effectiveness of high-dose megestrol in treating patients with metastatic breast cancer, endometrial cancer, or mesothelioma which cannot be treated with surgery or radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the clinical effects of high-dose oral megestrol in improving regression rate and prolonging survival in patients with breast or endometrial carcinoma or mesothelioma. II. Evaluate the immune, endocrine, and clinical effects of this regimen, with particular attention to effects on cachexia.

OUTLINE: This is a randomized study. Patients are stratified by performance status, dominant site of disease, and prior treatment with megestrol. Breast cancer patients are randomized to one of 3 doses of oral megestrol (800, 1,280, or 1,600 mg/day, divided qid). Female patients with other tumor types are nonrandomly assigned to receive oral megestrol at 1,600 mg/day. Male patients are nonrandomly assigned to a dose-finding study of megestrol. The first patient cohort receives megestrol at 480 mg/day in 3 divided doses, with further escalation for subsequent cohorts as tolerated. All patients continue therapy for at least 8 weeks, with treatment discontinued upon progression. Measurable lesions are evaluated every 2 months.

PROJECTED ACCRUAL: 9 evaluable breast cancer patients at each dose level will be entered; 14 patients will be required for each of the other disease categories. (As of 11/92, the study is temporarily closed to patients with prostate cancer.)

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented metastatic breast or endometrial carcinoma or mesothelioma not amenable to surgical and/or radiotherapeutic cure or long-term control Measurable soft tissue, bony, or visceral lesions required Indicator lesions other than blastic bony metastases and pleural effusions required for breast cancer Hormone receptor status (breast cancer): Estrogen-receptor-positive and/or progesterone-receptor-positive

PATIENT CHARACTERISTICS: Age: At least 18 Sex (breast cancer): Not specified Menopausal status (breast cancer): Any status Performance status: Not specified Life expectancy: At least 3 months Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since therapy Chemotherapy: At least 4 weeks since therapy Endocrine therapy: Breast cancer: At least disease stabilization achieved following tamoxifen or other hormonal manipulation if such treatment given previously At least 4 weeks since therapy Nonbreast cancer patients may be entered immediately after conventional doses of megestrol or other hormones Radiotherapy: At least 4 weeks since therapy Concomitant radiotherapy to nonindicator lesions allowed Surgery: At least 4 weeks since therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1987-12

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Wiseman, MD, FACP, Study Chair
Locations (1):
- St. Vincent Medical Center - Los Angeles, Los Angeles, California, United States